CLINICAL TRIAL: NCT04197037
Title: Prevalence Study of Sialorrhea in Inpatients and Outpatients Treated With Clozapine
Brief Title: Prevalence of Sialorrhea in Patients Treated With Clozapine
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Alicia Valiente, Professor, Parc de Salut Mar
Other Study IDs: 2019/8197
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Sialorrhea; Clozapine Adverse Reaction; Quality of Life
Keywords: Schizophrenia; Sialorrhea; Quality of life; Prevalence
MeSH Terms: conditions — Sialorrhea; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with schizophrenia treated with clozapine: People more than 18 with diagnosis of schizophrenia and treated with clozapine in a stable dose and stable status of the disease (at least 2-3 weeks).
  Interventions: Procedure: Evaluation of sialorrhea through questionnaires that measure daytime and nighttime sialorrhea and the impact on quality of life.

INTERVENTIONS:
Procedure: Evaluation of sialorrhea through questionnaires that measure daytime and nighttime sialorrhea and the impact on quality of life. — Sialorrhea will be evaluated by the Nocturnal hypersalivation rating scale (NHRS) and Drooling Severity and Frequency Scale (DSFS)

SUMMARY:
Clozapine is the "gold standard" antipsychotic drug for the treatment of resistant schizophrenia or resistant psychosis. Despite the high rates of good clinical response, the potential side effects can limit its use. Sialorrhea or excessive salivation is a side effect that occurs in 30-80% of people who receive this treatment and it can cause a decrease in self-esteem and feeling of security, greater social isolation and increase stigma.

The main objective of this study is to measure the prevalence of sialorrhea in inpatients and outpatients treated with clozapine and its consequences on the quality of life of people who are receiving this treatment.

A total of 129 patients over 18 years of age in treatment with clozapine will be recruited from different units of the Institute of Neuropsychiatry and Addictions (INAD) of the Parc de Salut Mar.

Sialorrhea will be evaluated by the nursing team with the Nocturnal Hypersalivation Rating Scale (NHRS), the Scale of Frequency and severity of salivation and the scale of impact on the quality of life. Also sociodemographic variables such as age, date of birth, race, date of diagnosis and clinical variables such as diagnosis, dose of clozapine and other treatments prescribed will be collected.

DETAILED DESCRIPTION:
BACKGROUND:

Clozapine is an atypical antipsychotic drug considered the "gold standard" in the treatment of resistant psychosis and also in patients who have had adverse effects with others drugs previously indicated as first line. It has been described that almost two thirds of patients who do not respond to first and second generation antipsychotics respond to clozapine treatment. Despite its effectiveness in positive, negative symptoms and the risk of suicide, clozapine presents a risk of adverse effects ranging from potentially dangerous ones. such as agranulocytosis or myocarditis, to others that are considered mild but that they can compromise the quality of life of patients and non-compliance. One of these mild, but extremely annoying, side effects is sialorrhea. The prevalence of sialorrhea secondary to clozapine reported by different studies range from 30% to 80% and it seems to be a dose-dependent relationship. This great variability observed in the studies probably has to do with the tendency that clinicians have to underestimate this side effect. In addition, the presence of sialorrhea can impact negatively in the subject causing a decrease in self-esteem and feeling of security, greater social isolation and an increase in stigma.

JUSTIFICATION OF THE STUDY:

Due to the consequences that sialorrhea has on the quality of life perceived by people in Clozapine treatment and the relationship with possible therapeutic abandonment, in addition to the low systematic evaluation of this side effect, it is considered relevant to establish a systematic evaluation of clozapine induced sialorrhea in the different mental health devices of our center.

OBJECTIVES:

To measure the prevalence of sialorrhea in patients treated with clozapine and its impact on subjective perception of quality of life. The possible relationship between the Clozapine dose and sialorrhea severity, as well as severity prediction will be evaluated based on the clinical and sociodemographic variables collected.

HYPOTHESIS:

1. The prevalence of sialorrhea in people treated with clozapine is at least 30% of patients receiving this antipsychotic treatment.
2. The presence of sialorrhea is directly related to a worse perception of the perceived quality of life in patients treated with clozapine.
3. The presence of sialorrhea is directly related to the prescribed dose of clozapine, presenting a dose-dependence relationship.
4. There is an association between the total daily dose of clozapine and the severity of sialorrhea in patients treated with clozapine.

MATERIAL AND METHODS:

Study design:

A quasi-experimental study will be carried out to measure the prevalence of sialorrhea in patients treated with clozapine in different Units of the INAD.

To estimate the sample size, people with the diagnosis of schizophrenia or schizoaffective disorder will be collected in the Units above mentioned in 2018, it was a sample size of 250.

Based on that the incidence of refractory schizophrenia is around 30% to 50% of cases, the number of patients potentially candidates to be treated with clozapine would be 125.

The final sample size has been calculated with the following tool available on the web http://.fisterra.com/mbe/investia/9samples/9samples.asp, with a 95% confidence interval and an accuracy of 3%, expecting sialorrhea in 30% of the cases and including a proportion of losses around 15%. The final sample will be 129 patients.

Methodology:

Nursing team will be responsible to inform the patients about the study, to enroll them and to obtain informed consent. Also they will administer 3 clinical scales previously used in hypersalivation studies (Maher et al. 2016; Wai Hong Man, Jantine Colen-de Koning, Peter Schulte and Ingrid van Haelst 2017) through the direct observation of the sialorrhea presented by the patient with stable treatment with clozapine. The scales will be administered only once and there won't be any longitudinal follow-up.

The scales are:

1. The Nocturnal Hypersalivation Rating Scale (NHRS): A validated scale of 5 items used to assess the severity of nocturnal salivation. Scores range from the non-presence of nocturnal salivation to wake up a minimum of 3 times during the night due to hypersalivation (Spivak et al. 1997).
2. Drooling Severity and Frequency Scale (DSFS): A validated scale to evaluate the severity of daytime sialorrhea (Rashnoo and Daniel 2015). Scores range from no presence of sialorrhea to a profuse sialorrhea where saliva wets the body or even objects and furniture (saliva falls on the table when the person is sitting) based on a 5-point scale.

   Both severity and frequency scores are added to give a final score of the daytime sialorrhea.
3. Impact on the quality of life scale: It is a 5-point scale that range from no impact on quality of life to a major problem.

In addition, sociodemographic variables such as age, date of birth, race, date of diagnosis, as well as variables clinics such as diagnosis, years of disease evolution, total daily dose of Clozapine treatment and other prescribed treatments.

All this information will be included in an anonymous database (subjects will be identified by a study code and the database will not include personal data).

Statistic analysis:

The data analysis will be carried out using the Statistical Package for the Social Sciences (SPSS statistical program), version 25.0. The distribution of the sociodemographic and clinical characteristics of the sample will be analyzed using descriptive statistics. Likewise, to describe the possible linear associations between quantitative variables related to clozapine and sialorrhea will use the coefficient of correlation. Finally, an exploratory regression analysis will be done to predict the severity of the sialorrhea based on clinical and sociodemographic variables. The limitations of the study will be the foreseeable studies of quasi-experimental studies: that do not allow establishing cause-effect relationships between variables or calculate incidence.

ELIGIBILITY:
Inclusion Criteria:

* People over 18 years
* In- and outpatients from different INAD Units
* Clozapine treatment with a stable dose (minimum one month without dose changes)

Exclusion Criteria:

* People under 18 years
* People receiving antipsychotic treatment other than clozapine (even though they present sialorrhea due to this treatment).
* It will not be exclusion criteria to be in treatment with other antipsychotics in conjunction with clozapine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of 129 patients over 18 years, treated with a stable dose of clozapine, will be selected through different units of the Institute of Neuropsychiatry and Addictions (INAD) of the Parc de Salut Mar.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of nocturnal sialorrhea in patients treated with clozapine | 1 week
  Prevalence of sialorrhea measured by Nocturnal hypersalivation rating scale. The values range from 0 to 4, the higher the score the greater the severity.
Prevalence of sialorrhea in patients treated with clozapine | 1 week
  Prevalence of daytime sialorrhea measured by Drooling Severity and Frequency Scale. The scale has two parts: one measures severity between 0-5 and the other measure frequency between 1-4. The higher the score, the more severe it is.

SECONDARY OUTCOMES:
Decrease in quality of life due to hypersalivation | 1 week
  Negative impact on quality of life due to hypersalivation measured by quality of life rating scale.The scale range is between 0 and 4, the higher the score the more severe it is.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Forum Parc de Salut Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Essali A, Al-Haj Haasan N, Li C, Rathbone J. Clozapine versus typical neuroleptic medication for schizophrenia. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD000059. doi: 10.1002/14651858.CD000059.pub2. PMID 19160174
- [Background] Maher S, Cunningham A, O'Callaghan N, Byrne F, Mc Donald C, McInerney S, Hallahan B. Clozapine-induced hypersalivation: an estimate of prevalence, severity and impact on quality of life. Ther Adv Psychopharmacol. 2016 Jun;6(3):178-84. doi: 10.1177/2045125316641019. Epub 2016 Mar 30. PMID 27354906
- [Background] Rashnoo P, Daniel SJ. Drooling quantification: Correlation of different techniques. Int J Pediatr Otorhinolaryngol. 2015 Aug;79(8):1201-5. doi: 10.1016/j.ijporl.2015.05.010. Epub 2015 May 18. PMID 26092552
- [Background] Remington G, Lee J, Agid O, Takeuchi H, Foussias G, Hahn M, Fervaha G, Burton L, Powell V. Clozapine's critical role in treatment resistant schizophrenia: ensuring both safety and use. Expert Opin Drug Saf. 2016 Sep;15(9):1193-203. doi: 10.1080/14740338.2016.1191468. Epub 2016 Jun 1. PMID 27207070
- [Background] Sockalingam S, Shammi C, Remington G. Clozapine-induced hypersalivation: a review of treatment strategies. Can J Psychiatry. 2007 Jun;52(6):377-84. doi: 10.1177/070674370705200607. PMID 17696024
- [Background] Spivak B, Adlersberg S, Rosen L, Gonen N, Mester R, Weizman A. Trihexyphenidyl treatment of clozapine-induced hypersalivation. Int Clin Psychopharmacol. 1997 Jul;12(4):213-5. doi: 10.1097/00004850-199707000-00005. PMID 9347382
- [Background] Syed R, Au K, Cahill C, Duggan L, He Y, Udu V, Xia J. Pharmacological interventions for clozapine-induced hypersalivation. Cochrane Database Syst Rev. 2008 Jul 16;2008(3):CD005579. doi: 10.1002/14651858.CD005579.pub2. PMID 18646130
- [Background] Man WH, Colen-de Koning J, Schulte P, Cahn W, van Haelst I, Heerdink E, Wilting I. Clozapine-induced hypersalivation: the association between quantification, perceived burden and treatment satisfaction reported by patients. Ther Adv Psychopharmacol. 2017 Sep;7(8-9):209-210. doi: 10.1177/2045125317707746. Epub 2017 May 1. No abstract available. PMID 28959433
- [Background] Yusufi B, Mukherjee S, Flanagan R, Paton C, Dunn G, Page E, Barnes TR. Prevalence and nature of side effects during clozapine maintenance treatment and the relationship with clozapine dose and plasma concentration. Int Clin Psychopharmacol. 2007 Jul;22(4):238-43. doi: 10.1097/YIC.0b013e32819f8f17. PMID 17519648
- [Derived] Sanagustin D, Martin-Subero M, Hogg B, Fortea L, Gardoki I, Guinart D, Roldan M, Angelats M, Cerro L, Navas D, Jimenez JD, Ortiz L, Ros R, Polo X, Ventura Y, Contreras J, Moreno-Alcazar A, Perez-Sola V, Amann BL, Valiente-Gomez A. Prevalence of clozapine-induced sialorrhea and its effect on quality of life. Psychopharmacology (Berl). 2023 Jan;240(1):203-211. doi: 10.1007/s00213-022-06294-3. Epub 2022 Dec 20. PMID 36538098
- See also: National Institute of Health and Clinical Excellence (NICE). 2014. "Psychosis and Schizophrenia in Adults." The NICE guidelines on treatment and management (February): 74-80. — http://www.nice.org.uk/guidance/cg178/evidence/full-guideline-490503565